CLINICAL TRIAL: NCT04028765
Title: POM PROM: Pitocin or Oral Misoprostol for PROM IOL in Nulliparous Women With Unfavorable Cervical Exams
Brief Title: Pitocin or Oral Misoprostol for PROM IOL
Acronym: POM PROM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Lisa Levine, Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 833536
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: PROM
MeSH Terms: interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oral Misoprostol (Active Comparator)
  Interventions: Drug: Misoprostol
- Oxytocin (Active Comparator)
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Misoprostol — Oral misoprostol 50 mcg every 4 hours for up to 6 doses or until cervical ripening is no longer indicated
  Arms: Oral Misoprostol
Drug: Oxytocin — IV Oxytocin 2 milliunits (mU)/min, increased by 2mU/min q15 minutes per hospital protocol
  Arms: Oxytocin

SUMMARY:
Premature rupture of membranes (PROM) is a common occurrence of pregnancies at term. A delay from PROM to labor is associated with an increased risk of intrauterine infection and associated maternal and fetal morbidity; therefore, induction of labor (IOL) is recommended. The ideal agent for IOL is not known, particularly among specific subpopulations. The primary aim of this study is to determine if oxytocin (Pitocin) or oral misoprostol results in a shorter interval to delivery after the start of induction among nulliparous women with unfavorable cervical exams with term PROM.

DETAILED DESCRIPTION:
Premature rupture of membranes (PROM) occurs in approximately 8% of pregnancies at term.1 Although onset of spontaneous labor is often prompt after membrane rupture, a delay from PROM to labor is associated with an increased risk of intrauterine infection and its associated maternal and fetal complications. For this reason, the American College of Obstetricians and Gynecologists (ACOG) endorses induction of labor for PROM "if spontaneous labor does not occur near the time of presentation."

The optimal method for PROM induction is less clear. Prior literature has examined the use of Pitocin (Oxytocin), vaginal and oral misoprostol, and dinoprost with mixed results. The TermPROM study found an increased risk of chorioamnionitis and Neonatal Intensive Care Unit (NICU) admission among women treated with vaginal misoprostol for induction.

The postulated link between vaginal misoprostol and chorioamnionitis is the need for vaginal examination for placement of the misoprostol; more vaginal examinations could potentially increase the risk for infection. Utilizing oral misoprostol would eliminate the need for a vaginal exam for administration, thereby potentially mitigating this risk of infection. Currently, vaginal and oral misoprostol as well as oxytocin are used routinely in clinical care based on provider discretion.

Among 7 randomized controlled trials examining the use of oral misoprostol as compared to oxytocin, two found oral misoprostol to result in faster induction to delivery, two found oxytocin to result in faster deliveries, and the remaining three found no difference between the two.3-9 These studies are limited by small sample size, inadequate reporting of patient demographics, varied misoprostol and oxytocin protocols, and inconsistent primary outcomes. Therefore, the utility of oral misoprostol in this population has not been established. Furthermore, its efficacy in specific patient populations is unreported in the literature.

The primary aim of this study is to determine if oxytocin or oral misoprostol results in a shorter interval to delivery after the start of induction among nulliparous women with unfavorable cervical exams with PROM.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* PROM </= 24 hours with no evidence of labor
* >/= 36 weeks gestation
* Agreeable to induction of labor
* Nulliparous
* Singleton pregnancy
* Vertex presentation
* Cervical dilation </=2 cm AND Bishop score < 8

Exclusion Criteria:

* Prior cesarean section
* Other contraindication to vaginal delivery
* Intrauterine Fetal Demise
* Major Congenital Anomaly
* Intraamniotic infection diagnosed at time of admission
* 36 weeks - 36 weeks and 6 days with unknown Group B Strep (GBS) status

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-01-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin No. 188: Prelabor Rupture of Membranes. Obstet Gynecol. 2018 Jan;131(1):e1-e14. doi: 10.1097/AOG.0000000000002455. PMID 29266075
- [Background] Hannah ME, Ohlsson A, Farine D, Hewson SA, Hodnett ED, Myhr TL, Wang EE, Weston JA, Willan AR. Induction of labor compared with expectant management for prelabor rupture of the membranes at term. TERMPROM Study Group. N Engl J Med. 1996 Apr 18;334(16):1005-10. doi: 10.1056/NEJM199604183341601. PMID 8598837
- [Background] Al-Hussaini TK, Abdel-Aal SA, Youssef MA. Oral misoprostol vs. intravenous oxytocin for labor induction in women with prelabor rupture of membranes at term. Int J Gynaecol Obstet. 2003 Jul;82(1):73-5. doi: 10.1016/s0020-7292(03)00136-x. No abstract available. PMID 12834947
- [Background] Crane JM, Delaney T, Hutchens D. Oral misoprostol for premature rupture of membranes at term. Am J Obstet Gynecol. 2003 Sep;189(3):720-4. doi: 10.1067/s0002-9378(03)00768-3. PMID 14526301
- [Background] Butt KD, Bennett KA, Crane JM, Hutchens D, Young DC. Randomized comparison of oral misoprostol and oxytocin for labor induction in term prelabor membrane rupture. Obstet Gynecol. 1999 Dec;94(6):994-9. doi: 10.1016/s0029-7844(99)00423-8. PMID 10576189
- [Background] Ngai SW, Chan YM, Lam SW, Lao TT. Labour characteristics and uterine activity: misoprostol compared with oxytocin in women at term with prelabour rupture of the membranes. BJOG. 2000 Feb;107(2):222-7. doi: 10.1111/j.1471-0528.2000.tb11693.x. PMID 10688506
- [Background] Mozurkewich E, Horrocks J, Daley S, Von Oeyen P, Halvorson M, Johnson M, Zaretsky M, Tehranifar M, Bayer-Zwirello L, Robichaux A 3rd, Droste S, Turner G; MisoPROM study. The MisoPROM study: a multicenter randomized comparison of oral misoprostol and oxytocin for premature rupture of membranes at term. Am J Obstet Gynecol. 2003 Oct;189(4):1026-30. doi: 10.1067/s0002-9378(03)00845-7. PMID 14586349
- [Background] Mbaluka CM, Kamau K, Karanja JG, Mugo N. EFFECTIVENESS AND SAFETY OF 2-HOURLY 20 MCG ORAL MISOPROSTOL SOLUTION COMPARED TO STANDARD INTRAVENOUS OXYTOCIN IN LABOUR INDUCTION DUE TO PRE-LABOUR RUPTURE OF MEMBRANES AT TERM: A RANDOMISED CLINICAL TRIAL AT KENYATTA NATIONAL HOSPITAL. East Afr Med J. 2014 Sep;91(9):303-10. PMID 26866082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Began: August 2019 End: May 2023 (Last participant follow-up completed 1/8/2023. Additional subjects were screened/approached for participation through 5/2023.) Location: Labor and Delivery
Groups:
- Oxytocin: Oxytocin: IV Oxytocin 2 milliunits (mU)/min, increased by 2mU/min q15 minutes per hospital protocol. Max 40 mU/min
Period: Overall Study
Arm/Group | Oral Misoprostol | Oxytocin
Started | 52 | 56
Completed | 52 | 56
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Misoprostol | Oxytocin | Total
Number analyzed (Participants) | 52 | 56 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (5.4) | 28.5 (5.9) | 29.2 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 56 | 108
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 27 | 25 | 52
  Race: White | 20 | 20 | 40
  Race: Asian | 4 | 6 | 10
  Race: Hispanic, not otherwise specified | 1 | 5 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 56 | 108
Public Insurance [Count of Participants; unit: Participants] | 20 | 23 | 43
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 31.9 [26.7 to 37.1] | 31.9 [28.7 to 35.2] | 31.9 [27.6 to 36.2]
Prenatal Visit Number [Median (Inter-Quartile Range); unit: Visits] | 9 [7 to 10] | 9 [7 to 10] | 9 [7 to 10]
Gestational age at Rupture of Membranes [Median (Inter-Quartile Range); unit: Weeks] | 39.7 [38.9 to 40.5] | 39.3 [38.5 to 40.2] | 39.4 [38.6 to 40.3]
Starting Cervical Dilation [Mean (Standard Deviation); unit: Centimeters] | 1.1 (0.6) | 1.1 (0.5) | 1.1 (0.5)
Starting Bishop Score [Mean (Standard Deviation); unit: Units on a scale.] — The Bishop score is a commonly used method to rate cervical ripeness for induction of labor. The score ranges from 0-12 with points awarded for cervical dilation, cervical effacement, fetal station, cervical consistency, and cervical position. Scores for each of those 5 categories are added to generate a total score. Higher scores indicate more favorable (or ripe) cervical examinations
  Units on a scale. | 3.6 (1.5) | 3.9 (1.7) | 3.8 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Time From Induction of Labor (IOL) to Delivery
Description: Time (hours) from start of IOL (As defined by receipt of first medication for induction of labor) to delivery of infant.
Time Frame: Time (hours) from start of IOL (As defined by receipt of first medication for induction of labor) to delivery of infant.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Oral Misoprostol | Oxytocin
Number analyzed (Participants) | 52 | 56
Hours | 18.1 [12.2 to 24] | 14.9 [10.9 to 18.9]

2. Secondary Outcome: Infection
Description: Suspected intraamniotic infection
Time Frame: Enrollment to Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Misoprostol | Oxytocin
Number analyzed (Participants) | 52 | 56
Participants | 8 | 6

3. Secondary Outcome: Time From Premature Rupture of Membranes (PROM) to Delivery
Time Frame: Time (hours) from PROM (as reported by patient) to delivery of infant
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Oral Misoprostol | Oxytocin
Number analyzed (Participants) | 52 | 56
Hours | 25.8 [18.5 to 33.2] | 22.1 [17.3 to 26.9]

4. Secondary Outcome: Time From IOL to Vaginal Delivery
Time Frame: Time from IOL (as defined by receipt of first medication for induction) to vaginal delivery
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Oral Misoprostol | Oxytocin
Number analyzed (Participants) | 52 | 56
Hours | 17.9 [11.7 to 24.1] | 12.9 [9.2 to 16.4]

5. Secondary Outcome: Time From PROM to Vaginal Delivery
Time Frame: Time (hours) from PROM (as reported by patient) to vaginal delivery
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Oral Misoprostol | Oxytocin
Number analyzed (Participants) | 52 | 56
Hours | 24.9 [16.9 to 32.9] | 21.6 [17.4 to 25.8]

6. Secondary Outcome: Cesarean Delivery
Description: Cesarean section rate
Time Frame: Enrollment to Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Misoprostol | Oxytocin
Number analyzed (Participants) | 52 | 56
Participants | 13 | 14

7. Secondary Outcome: Maternal Morbidity
Description: Composite maternal morbidity: postpartum hemorrhage, blood transfusion, endometritis, wound infection, venous thromboembolism (VTE), hysterectomy, Intensive care unit (ICU) admission, readmission within 4 weeks, death
Time Frame: Enrollment to 4 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Misoprostol | Oxytocin
Number analyzed (Participants) | 52 | 56
Participants | 8 | 9

8. Secondary Outcome: Neonatal Morbidity
Description: Composite neonatal morbidity: NICU admission > 48 hours, neonatal blood transfusion, hypoxic ischemic encephalopathy, intraventricular hemorrhage grade III or IV, headcooling, severe respiratory distress syndrome, necrotizing enterocolitis, sepsis, death
Time Frame: Enrollment to hospital discharge (On average 2-4 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Misoprostol | Oxytocin
Number analyzed (Participants) | 52 | 56
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: From trial enrollment to one month post-delivery (Maternal) or hospital discharge (Neonatal)
Description: Adverse events as described per maternal and neonatal subject. Described adverse event numbers are per event (ie. subject may have experienced more than one event).
Groups:
- Oral Misoprostol-Mothers: Misoprostol: Oral misoprostol 50 mcg every 4 hours for up to 6 doses or until cervical ripening is no longer indicated Adverse Maternal Events Only
- Oxytocin-Mothers: Oxytocin: IV Oxytocin 2 milliunits (mU)/min, increased by 2mU/min q15 minutes per hospital protocol. Max 40 mU/min Adverse Maternal Events only
- Oral Misoprostol-Fetus/Neonate: Misoprostol: Oral misoprostol 50 mcg every 4 hours for up to 6 doses or until cervical ripening is no longer indicated Adverse Neonatal Events Only
- Oxytocin-Fetus/Neonate: Oxytocin: IV Oxytocin 2 milliunits (mU)/min, increased by 2mU/min q15 minutes per hospital protocol. Max 40 mU/min Adverse Neonatal Events only
Arm/Group | Oral Misoprostol-Mothers | Oxytocin-Mothers | Oral Misoprostol-Fetus/Neonate | Oxytocin-Fetus/Neonate
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/56 | 0/52 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/56 | 1/52 | 0/56
Other Adverse Events (participants affected / at risk) | 3/52 | 3/56 | 1/52 | 2/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Misoprostol-Mothers (N=52) | Oxytocin-Mothers (N=56) | Oral Misoprostol-Fetus/Neonate (N=52) | Oxytocin-Fetus/Neonate (N=56)
Neonatal Hypoxic Ischemic Encephalopathy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Oral Misoprostol-Mothers (N=52) | Oxytocin-Mothers (N=56) | Oral Misoprostol-Fetus/Neonate (N=52) | Oxytocin-Fetus/Neonate (N=56)
NICU Admission > 48 hours (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 0/0 (0) | 1 (1) | 2 (2)
Postpartum Readmission (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0/0 | 0/0
Blood transfusion (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/65/NCT04028765/Prot_SAP_002.pdf
  • Informed Consent Form (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT04028765/ICF_003.pdf